CLINICAL TRIAL: NCT06444789
Title: AI-based Parkinson's Disease Risk Assessment and Prognosis - Digital Biomarkers Development, Validation and Verification Study (AI-PROGNOSIS dBM-DEV Study)
Brief Title: AI-PROGNOSIS - Digital Biomarkers Development Study (dBM-DEV)
Acronym: dBM-DEV
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: European Union (Other); University Hospital Carl Gustav Carus (Other); Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0184 - RC31/24/0031
Record Dates: First submitted 2024-05-14; First posted 2024-06-06 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
Keywords: REM sleep behaviour disorder
MeSH Terms: conditions — Parkinson Disease; REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Development cohort of patients with known RBD: Detection of RBD signs by using the connected smartwach during 4 weeks
  Interventions: Device: connected smartwatch
- Development cohort of matched controls = people who don't have RBD age and sex matched: Detection of RBD signs by using the connected smartwach during 4 weeks
  Interventions: Device: connected smartwatch
- Confirmation cohort of parkinson disease patients = people who are supposed to have RBD: Detection of RBD signs by using the connected smartwach during 3 months
  Interventions: Device: connected smartwatch

INTERVENTIONS:
Device: connected smartwatch — The smartwatch is worn by the patient and data are sent automatically to a server that detects if there are signs of RBD.

SUMMARY:
dBM-dev study is a multicentre low-intervention research study which concerns REM sleep behaviour disorder (RBD) who is the best predictor for neurodegenerative diseases including Parkinson's disease (PD). RBD can only be confirmed by polysomnography, which is a cumbersome procedure. The main objective of this study is to identify a novel, robust dBM for the detection of RBD using smartwatch-based recordings of passive data.The study is conducted step-wise on two subsequent cohorts referred to as the development cohort and the confirmation cohort.

DETAILED DESCRIPTION:
The development cohort comprises 30 patients with RBD and 30 matched controls on sex and age with patients RBD.

The confirmation cohort comprises 30 patients with PD. Following a baseline visit comprising standard clinical evaluation and Parkinson questionnaires, participants will undergo daily-life dBM tracking over a duration of 4 weeks for development cohort and 3 months for confirmation cohort. Additionally, PD patients enrolled in the confirmation cohort will receive a polysomnography which permits to verificate if they have a RBD. The investigation is conducted in four European sites.

ELIGIBILITY:
Inclusion Criteria for development cohort:

Group of RBD patients

* Diagnosis of RBD (confirmed by polysomnography)
* Able to use a compatible smartphone with the study app
* Having a care partner with whom they share their bedroom at night

Group of Healthy matched controls:

* Healthy volunteers age and sex matched to the enrolled RBD patients.
* Able to use a compatible smartphone with the study app
* No history of RBD.

Inclusion Criteria for confirmation cohort

* Clinical confirmed diagnosis of PD
* RBD Screening Questionnaire score : 3 - 12 points
* Absence of dementia
* Able to use a compatible smartphone with the study app
* Having a care partner with whom they share their bedroom at night

Exclusion Criteria for all cohorts:

Inability to consent for study procedures as judged by the investigator. Lacking motivation to participate in study procedures as judged by the investigator.

Lack of social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1 group of persons with RBD
  1 group of persons without RBD
  1 group of persons with Parkinson disease
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2024-09-20 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of nights in a confirmation cohort in which RBD episodes are indicated by a score (digital biomarker) derived from passive actigraphy and photoplethysmography data captured by a smartwatch | 4 weeks
  the digital biomarker will be identified from passive actigraphy and photoplethysmography data of a separate development cohort

SECONDARY OUTCOMES:
correlation between a) and b) | 4 weeks for a) 3 months for b)
  1. the incidence of daytime somnolence episodes per week indicated by a score (digital biomarker) derived from passive actigraphy and photoplethysmography data captured by a smartwatch. The digital biomarker will be identified from passive actigraphy and photoplethysmography data of a separate development cohort
  2. the score of the Epworth Sleepiness Scale at baseline, measured by the Spearman correlation coefficient, in a confirmation cohort
Number of camera-based movement assessments acquired by each participant relative to the number of scheduled camera-based movement assessments. | 4 weeks (for development cohort) and 3 months (for confirmation cohort)
Number of cognitive tasks completed by each participant relative to the number of scheduled cognitive tasks. | 4 weeks (for development cohort) and 3 months (for confirmation cohort)

CONTACTS AND LOCATIONS:
Overall Officials: Margherita FABBRI, Principal Investigator — Toulouse Hospital; Björn FALKENBURGER, Study Chair — University Hospital Carl Gustav Carus of Dresden
Locations (4):
- Neurology Toulouse Hospital, Toulouse, France
- Klinik und Poliklinik für Neurologie of University Hospital (Regulatory autorization pending), Dresden, Germany
- Hospital Ruber Internacional, Madrid, Spain
- King's college of London (Regulatory authorization pending), London, United Kingdom

REFERENCES:
- See also: Related Info — https://www.ai-prognosis.eu